CLINICAL TRIAL: NCT04170387
Title: Passive Movements of Fingers and Impact on Cognitive Impairment and Blurry Mind in Fibromyalgic Patients: Exploratory Study
Brief Title: Can a Relaxometer Improve Cognitive Impairment of Fibromyalgia Patients
Acronym: Fibrorilax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Fibrorilax
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia Syndrome; Fibromyalgia; Pain, Chronic; Impairment; Cognitive Impairment
Keywords: Relaxometer; Mini Mental State Examination; Fibromyalgia Impact Questionnaire; Cognitive Impairment; Rehabilitation; Fingers
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Cognitive Dysfunction | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: Two cohorts of 20 patients each. The first group includes patients affected by fibromyalgia and the other is the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxometer fibromyalgia cases (Experimental): Repetition 6 minutes pre-set programme with the relaxometer 60 seconds 34 movements/minute 3 seconds 55 movements/minute 60 seconds 34 movements/minute 60 seconds 55 movements/minute 90 seconds 34 movements/minute 5 seconds 55 movements/minute 90 seconds 34 movements/minute
  Interventions: Other: Relaxometer
- Relaxometer controls (Active Comparator): Repetition 6 minutes pre-set programme with the relaxometer 60 seconds 34 movements/minute 3 seconds 55 movements/minute 60 seconds 34 movements/minute 60 seconds 55 movements/minute 90 seconds 34 movements/minute 5 seconds 55 movements/minute 90 seconds 34 movements/minute
  Interventions: Other: Relaxometer

INTERVENTIONS:
Other: Relaxometer — Day 1: signing of informed consent, medical history, physical examination, Mini-Mental State Examination (MMSE), Fibromyalgia Impairment Questionnaire revised (FIQ-R), repetition of 6 minutes relaxometer pre-set programme for 3 times Day 2: repetition of 6 minutes relaxometer pre-set programme for 3 times Day 3: repetition of 6 minutes relaxometer pre-set programme for 3 times Day 8: 6 minutes relaxometer pre-set programme once Day 10: 6 minutes relaxometer pre-set programme once, Mini-Mental State Examination Day 30: Mini-Mental State Examination (MMSE), Fibromyalgia Impairment Questionnaire revised (FIQ-R)
  Other Names: Mini-Mental State Examination (MMSE); Fibromyalgia Impairment Questionnaire revised (FIQ-R)

SUMMARY:
The aim of the study is to evaluate the differences in cognitive performance and quality of life, after a cycle of treatment with the relaxometer, between a group of patients affected by fibromyalgia and a control group.

DETAILED DESCRIPTION:
The relaxometer is a device designed for the physical rehabilitation of patients with functional problems of upper limbs. It works by moving passively the patient's fingers in a gradual way (with different speeds) in all directions of space, which is innovative compared to similar machines already on the market.

The device consists of an electrical supply unit and two handling units made of 10 silicone tips of different sizes for the placement of fingers and it works with a six-minute pre-set program. It has obtained patent and certification mark and it has been used in the rehabilitation of patients with joint stiffness induced by specific working activities, as musicians.

After the treatment these patients reported a remarkable improvement of motor skills and articulation of fingers, in addition to a parallel improvement of cognitive abilities such as concentration, visual acuity and mnemonic learning.

In sight of this, the aim of the study is to establish whether the application of this treatment in a small group patients affected by fibromyalgia and cognitive impairment is able to improve some aspects of the cognitive dysfunction measured with appropriate functional tests and comparing the results with a control group of patients not affected by this condition.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgic Syndrome diagnosed according to the criteria of American College of Rheumatology 2016 (ACR 2016)
* moderate-severe cognitive impairment according to the Symptoms Severity Score (SS)
* informed consent gathered

Exclusion Criteria:

* contraindication to passive handling of fingers (severe arthritis, fractures or unconsolidated traumatic outcomes, not healed wounds, finger amputations, contact allergies to substances contained in the relaxometer)
* informed consent not gathered
* drug addiction
* brain stroke

Withdrawal from study

* withdrawal of informed consent
* treatment non completed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-10-14 (Estimated)

PRIMARY OUTCOMES:
Assessment of differences in cognitive performance of patients affected by fibromyalgia with cognitive impairment before and after a cycle of treatment with the relaxometer. | 4 weeks
  Mini-Mental State Examination (MMSE) administered before the first treatment with the relaxometer (T0), after the last treatment with the relaxometer (T1, on the 10^ day from the first treatment) and on the 30^ day from the first treatment (T2).
  Mini-Mental State Examination is a 30 point questionnaire used to measure cognitive impairment.
  Normal cognition 24-30 points Mild cognitive impairment 19-23 points Moderate cognitive impairment 10-18 points Severe cognitive impairment <9 points The score is corrected for educational attainment and age, according to MMSE guidelines.

SECONDARY OUTCOMES:
Evaluate the differences in cognitive performance obtained at the end of treatment, between the case group (patients affected by fibromyalgia with cognitive impairment) and the control group. | 52 weeks
  Comparison of Mini-Mental State Examination (MMSE) results.
  Mini-Mental State Examination is a 30 point questionnaire used to measure cognitive impairment.
  Normal cognition 24-30 points Mild cognitive impairment 19-23 points Moderate cognitive impairment 10-18 points Severe cognitive impairment <9 points The score is corrected for educational attainment and age, according to MMSE guidelines.
Evaluate the differences in quality of life (QoL) of patients affected by fibromyalgia before and after a cycle of treatment with the relaxometer, comparing them with the control group. | 52 weeks
  Fibromyalgia Impact Questionnaire revised (FIQ-R) administered before the first treatment with the relaxometer and during the last examination on the 30^ day from the first treatment.
  Fibromyalgia Impact Questionnaire revised (FIQ-R) explores three domains: function, overall impact, and symptoms. The score of each domain is divided by a specific number
  * Function domain sum (0-90) divided by 3 (upper limit 30)
  * Overall impact domain sum (0-20) divided by one (0-20)
  * Symptom domain sum (0-100) divided by 2 (upper limit 50) The three resulting domain scores are added together to obtain the total score of the Fibromyalgia Impact Questionnaire revised (FIQ-R) range 0-100.
  75-100 Extreme fibromyalgia 60-74 Severe fibromyalgia 43-59 Moderate fibromyalgia 0-42 Mild fibromyalgia

IPD SHARING:
Plan to Share IPD: No